CLINICAL TRIAL: NCT04384159
Title: Transient Versus Bidimensional Shear Wave Elastography in Serial Combination Strategy to Diagnose Advanced Fibrosis in NAFLD Patients
Brief Title: Combination Diagnostic Strategies in NAFLD
Acronym: CombinationSSI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0281
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Chronic Liver Disease
Keywords: Liver elastography; Liver fibrosis; Non-invasive diagnosis; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serial combination of biological and elastography tests is accurate to diagnosing advanced fibrosis in non-alcoholic fatty liver disease (NAFLD) patients. In this study, the investigators compared the diagnostic performances of a 2-step strategy using either vibration-controlled transient elastography (VCTE) or bidimensional shear wave elastography with Supersonic imagine (2D-SWE-SSI), and analysed the added-value of a 3-step strategy.

DETAILED DESCRIPTION:
The investigators retrospectively selected all consecutive adult patients with suspicion of NAFLD who had undergone liver biopsy from November 2011 to July 2019 in 2 French academic centers, Angers and Bordeaux university hospitals. A total of 577 patients were included. Among them, 291 had been previously included in a prospective study comparing diagnostic performances of several non-invasive tests in NAFLD patients. Inclusion criteria were: Age≥18yo, 2D-SWE-SSI and VCTE performed within the two weeks prior to liver biopsy. Exclusion criteria were high alcohol consumption (i.e., >21 drinks, on average, per week in men and >14 drinks, on average, per week in women), associated causes of liver disease (alcoholic, viral, or other causes of liver injury), other aetiologies than NAFLD on pathological examination, and a liver biopsy length of less than 10 mm and/or fewer than 6 portal spaces and/or more than 2 fragments, except for in cases of cirrhosis.

ELIGIBILITY:
Inclusion criteria:

- PAtients who underwent a liver biopsy for a suspicion of NAFLD, and liver stiffness evaluation with either Fiborscan and Bidimensional shear wave elastography

Exclusion criteria:

* Other aetiologies of chronic liver disease
* biopsy length under 10mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver biopsy for the diagnosis of a NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracyclassification | 1 day
  Diagnostic accuracyclassification

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Cassinotto, PU-PH, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC